CLINICAL TRIAL: NCT02950675
Title: The Relationship of Body Function, Participation and Quality of Life in Patients With Burn: A Longitudinal Study
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 104-9848B
Record Dates: First submitted 2016-10-10; First posted 2016-11-01 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2019-01

CONDITIONS: Burn
Keywords: Burn patient; Developmental Disabilities; Body function; Participation; Quality of Life; longitudinal study
MeSH Terms: conditions — Burns; Developmental Disabilities

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Normal Adult: Control:Normal Adult
- Burn Patient: The burn patient will be identified according to the diagnoses (ICD-9-CM code: 940-949).

SUMMARY:
The relationship of body function, participation and quality of life in patients with burn: A longitudinal study

DETAILED DESCRIPTION:
Early rehabilitation to partial-thickness and full-thickness dermal injury are of vital importance for burn patient. Literature reviews have shown that burn patients experiences ADL and quality of life (QOL) difficulties. Due to varied severity, the outcome and expression of each patient also differs. The limitation of body function may consequently affect social participation and QOL thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of burn injuries admitted to Burn Center or followed in burn clinic
* Age >14
* No mental diseases
* Understand written Chinese or could complete the questionnaires with staff's assistance

Exclusion Criteria:

* Died during or after hospitalization
* Refused to participate in the investigation
* Concurrent medical illness that affecting the subjectivity of post burn sequelae (ex. progressive muscular or mental diseases, trauma or seizure)
* Age >74

Ages: 14 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The investigators will have Normal Adult (n=30~40) and Burn Patient (n=80-90) from 14-74 years old under consent of their family.
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2016-07; Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Change in bodily function in baseline, 3 month, 12 month, 18 month, 24 month, 30 month and 36 month follow up | baseline, 3 month, 12 month, 18 month, 24 month, 30 month and 36 month
  Vancouver Scar Scale (VSS)

SECONDARY OUTCOMES:
Change in muscle strength change in baseline, 3 month, 12 month, 18 month, 24 month, 30 month and 36 month follow up | baseline, 3 month, 12 month, 18 month, 24 month, 30 month and 36 month
  MicroFET
Change in activities of daily living in baseline, 3 month, 12 month, 18 month, 24 month, 30 month and 36 month follow up | baseline, 3 month, 12 month, 18 month, 24 month, 30 month and 36 month
  Functional Independence Measure (FIM)
Change in individual independency in baseline, 3 month, 12 month, 18 month, 24 month, 30 month and 36 month follow up | baseline, 3 month, 12 month, 18 month, 24 month, 30 month and 36 month
  Manual for the Care and Needs Scale
Change in quality of life in baseline, 3 month, 12 month, 18 month, 24 month, 30 month and 36 month follow up | baseline, 3 month, 12 month, 18 month, 24 month, 30 month and 36 month
  The Burn-Specific Health Scale-Brief

CONTACTS AND LOCATIONS:
Overall Officials: Katie P Wu, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No